CLINICAL TRIAL: NCT07071012
Title: Effect of External Oblique Intercostal Block Versus Paravertebral Block on Postoperative Pain and Complications in Open Nephrectomy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Almıla Gulsun Pamuk, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-24040
Record Dates: First submitted 2025-07-06; First posted 2025-07-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nephrectomy; Pain Scores; Paravertebral Block; External Oblique Intercostal Block
Keywords: postoperative pain; nephrectomy; External oblique intercostal block; paravertebral block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Morphine; Acetaminophen; Diclofenac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block (Active Comparator): Patients scheduled to undergo thoracic paravertebral block will receive an injection of 20 ml of 0.25% bupivacaine hydrochloride into the paravertebral space between the parietal pleura and the costotransverse ligament using a block needle under ultrasound guidance.
  Interventions: Drug: Bupivacaine; Drug: morphine; Drug: paracetamol; Drug: Diclofenac
- External Oblique Intercostal Block (Active Comparator): Patients scheduled to undergo an external oblique intercostal block will receive an injection of 30 ml of 0.25% bupivacaine hydrochloride between the external oblique muscle and the intercostal muscle at the level of the 6th rib, using a block needle under ultrasound guidance.
  Interventions: Drug: Bupivacaine; Drug: morphine; Drug: paracetamol; Drug: Diclofenac

INTERVENTIONS:
Drug: Bupivacaine — Used for regional anesthesia during nephrectomy procedure (e.g., paravertebral or external oblique intercostal block)
Drug: morphine — Used for postoperative pain control via PCA device
Drug: paracetamol — Used as part of postoperative multimodal analgesia
Drug: Diclofenac — Administered for postoperative pain management

SUMMARY:
This study aims to compare the effects of external oblique intercostal block versus paravertebral block on postoperative pain and complications in patients undergoing open nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 90 years
* Stage 2 renal cell carcinoma scheduled for open radical nephrectomy without lymph node dissection
* ASA classification I-III
* Mini-Mental State Examination score ≥24
* Provided written informed consent

Exclusion Criteria:

* Neuropathy
* Hepatic failure
* Coagulopathy
* Local anesthetic allergy
* Mini-Mental State Examination score <24
* Refusal to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score | Up to 24 hours after surgery
  Pain intensity measured using Visual Analog Scale at rest and during movement (Visual Analog Scale ranging from 0 = no pain to 10 = worst pain imaginable; higher scores indicate worse pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Medicine Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No